CLINICAL TRIAL: NCT02352103
Title: The Impact of Retzius-sparing Approach for Robot-assisted Laparoscopic Radical Prostatectomy on Short-term Continence Recovery: Randomized Controlled Trial
Brief Title: Impact of Robot-assisted Radical Prostatectomy Technique on Short-term Continence Recovery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Mani Menon, Director, Vattikuti Urology Institute, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9220
Record Dates: First submitted 2015-01-22; First posted 2015-02-02 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Urinary Incontinence
Keywords: prostate cancer; Urinary continence; robotic assisted radical prostatectomy; Vattikuti Urology Institute (VIP) radical prostatectomy; Retzius sparing radical prostatectomy
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Active Comparator): Vattikuti Urology Institute radical prostatectomy da Vinci Surgical System
  Interventions: Procedure: Vattikuti Urology Institute radical prostatectomy; Device: da Vinci Surgical System
- Treatment arm (Experimental): Retzius sparing radical prostatectomy da Vinci Surgical System
  Interventions: Procedure: Retzius sparing radical prostatectomy; Device: da Vinci Surgical System

INTERVENTIONS:
Procedure: Retzius sparing radical prostatectomy — Robotic assisted laparoscopic radical prostatectomy based on Retzius sparing technique
  Arms: Treatment arm
Procedure: Vattikuti Urology Institute radical prostatectomy — Robotic assisted laparoscopic radical prostatectomy based on Vattikuti Urology Institute technique
  Arms: Control arm
Device: da Vinci Surgical System — The da Vinci Surgical System is a sophisticated robotic platform designed to expand the surgeon's capabilities and offer a state-of-the-art minimally invasive option for major surgery.

SUMMARY:
To assess and compare the short-term post-operative continence recovery rate in two cohorts of men undergoing Robot Assisted Radical Prostatectomy (RARP), each randomized to undergo RARP with Vattikuti Institute technique or Retzius sparing technique.

DETAILED DESCRIPTION:
Traditionally, RARP is performed using a trans-peritoneal technique that pass anteriorly to the bladder. This technique necessitates the dissection and/or manipulation of many structures, which might compromise post-operative urinary continence recovery. These structures include the pubo-prostatic ligament, Santorini plexus, neurovascular bundle, and veil of Aphrodite. Recently, a "Retzius-sparing" technique to perform RARP has beed described. This approach passes posteriorly to the bladder, through the space of Douglas, which should minimize the damaged to the aforementioned structure. Theoretically, the latter technique should improve post-operative urinary continence recovery. However, a randomized comparison between the "traditional" RARP and "Retzius-sparing" RARP is still lacking.

ELIGIBILITY:
Inclusion Criteria:

* All patients with newly diagnosed prostate cancer undergoing robotic-assisted radical prostatectomy at the Vattikuti Urology Institute (performed by single surgeon, MM) as the primary treatment modality
* Be able to read and speak English and be able to provide written informed consent

Exclusion Criteria:

* patients with high risk prostate cancer,defined as a biopsy Gleason score ≥8 and/or a pre-operative prostate specific antigen value ≥20 ng/ml.
* evidence of clinical nodal involvement (cN1) or metastatic disease (M1)
* patients participating in a competing study
* patients with pre-operative urinary incontinence.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mani Menon, MD, Principal Investigator — Henry Ford Hospital
Locations (2):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dalela D, Jeong W, Prasad MA, Sood A, Abdollah F, Diaz M, Karabon P, Sammon J, Jamil M, Baize B, Simone A, Menon M. A Pragmatic Randomized Controlled Trial Examining the Impact of the Retzius-sparing Approach on Early Urinary Continence Recovery After Robot-assisted Radical Prostatectomy. Eur Urol. 2017 Nov;72(5):677-685. doi: 10.1016/j.eururo.2017.04.029. Epub 2017 May 6. PMID 28483330
- [Result] Menon M, Dalela D, Jamil M, Diaz M, Tallman C, Abdollah F, Sood A, Lehtola L, Miller D, Jeong W. Functional Recovery, Oncologic Outcomes and Postoperative Complications after Robot-Assisted Radical Prostatectomy: An Evidence-Based Analysis Comparing the Retzius Sparing and Standard Approaches. J Urol. 2018 May;199(5):1210-1217. doi: 10.1016/j.juro.2017.11.115. Epub 2017 Dec 7. PMID 29225060
- See also: A Pragmatic Randomized Controlled Trial Examining the Impact of the Retzius-sparing Approach on Early Urinary Continence Recovery After Robot-assisted Radical Prostatectomy — https://pubmed.ncbi.nlm.nih.gov/28483330/
- See also: Functional Recovery, Oncologic Outcomes and Postoperative Complications after Robot-Assisted Radical Prostatectomy: An Evidence-Based Analysis Comparing the Retzius Sparing and Standard Approaches — https://pubmed.ncbi.nlm.nih.gov/29225060/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm | Treatment Arm
Started | 60 | 60
Completed | 60 | 59
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Treatment Arm | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.5 [56 to 67] | 61 [55 to 67] | 61 [56 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 60 | 60 | 120
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 28 [26.4 to 30.9] | 27.9 [26.1 to 30.6] | 28 [26.2 to 30.7]
preoperative prostate specific antigen level [Median (Inter-Quartile Range); unit: ng/ml] | 5.4 [3.7 to 7.3] | 5.7 [4.7 to 7.4] | 5.6 [4.1 to 7.3]
preoperative IPSS score [Median (Inter-Quartile Range); unit: units on a scale] — International Prostatic Symptom Score (IPSS) objectively assesses urinary symptoms. It ranges from 0 to 35, with higher scores indicating worse urinary symptoms
  units on a scale | 6.5 [3 to 13] | 7 [3 to 12] | 7 [3 to 12]
preoperative SHIM score [Median (Inter-Quartile Range); unit: units on a scale] — SHIM (Sexual Health Inventory for Men) objectively asses sexual function. It ranges from 0-25, with higher scores indicating better sexual function.
  units on a scale | 20 [8 to 25] | 20 [14 to 24] | 20 [11 to 25]
NCCN clinical risk [Count of Participants; unit: Participants] — NCCN (National Comprehensive Cancer Network) risk categorizes prostate cancer based on their likelihood of disease progression, recurrence and outcomes, into low, intermediate, high and very high risk groups. It uses clinical information (i.e information available PRIOR to surgery) for this (i.e PSA, biopsy gleason score and clinical T stage)
  Participants
    Low Risk | 15 | 14 | 29
    Intermediate Risk | 45 | 46 | 91

OUTCOME MEASURES:

1. Primary Outcome: Urinary Continence Recovery
Description: 24-hour pad weights
Time Frame: One week after the removal of the suprapubic urinary catheter
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 60 | 59
grams | 25 [3 to 133] | 5 [0 to 25]

2. Secondary Outcome: Number of Participants With Urinary Continence Recovery
Description: 0 pad per day
Time Frame: within 3 months from the intervention
Measure: Number; unit: participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 60 | 60
participants | 46 | 35

3. Secondary Outcome: Number of Participants With Peri and Postoperative Complications
Description: Clavien-Dindo complications
Time Frame: 1-year median follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 60 | 60
Participants | 7 | 11

4. Secondary Outcome: Number of Participants Who Regained Potency Postoperatively (as Measured by Sexual Health Inventory for Men (SHIM) Score of 17 or Greater)
Description: SHIM ranges from 0-25 with higher scores indicating better sexual function; a score of >=22 is normal and >=17 is considered mild ED
Time Frame: 1-year median follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 60 | 60
Participants | 27 | 26

5. Secondary Outcome: Number of Participants Who Had Biochemical Recurrence (Post-operative Prostate-Specific Antigen (PSA) Value >=0.2 ng/ml)
Description: Patients without biochemical evidence of disease recurrence (i.e. postop PSA >=0.2 ng/mL)
Time Frame: 1-year median follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 60 | 60
Participants | 56 | 50

6. Secondary Outcome: Post-operative Urinary Function and Urinary Function-related Quality of Life
Description: International Prostatic Symptom Score (continuous score from 0-35, higher scores indicating worse urinary function)
Time Frame: Within 3 months from the intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 60 | 60
score on a scale | 5.5 [4.3 to 6.7] | 4.4 [3.4 to 5.4]

7. Other Pre Specified Outcome: Number of Patients Who Regained Urinary Continence Postoperatively
Description: 0 pad per day
Time Frame: 1 year median follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 60 | 60
Participants | 53 | 58

8. Other Pre Specified Outcome: Post-operative Urinary Function and Urinary Function-related Quality of Life
Description: MSKCC (Memorial Sloan Kettering Cancer Center) STAR questionnaire (symptom tracking and reporting). Score ranges from 0-25, with higher scores indicating better urinary function
Time Frame: 1 year median follow up
Population: The numbers in this analyses are different from the primary analyses as some patients were lost to follow up (by one year)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 48 | 52
score on a scale | 20 [16 to 23] | 20 [17 to 24]

ADVERSE EVENTS:
Arm/Group | Control Arm | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 5/60 | 7/60
Other Adverse Events (participants affected / at risk) | 2/60 | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=60) | Treatment Arm (N=60)
Lymphocele (Blood and lymphatic system disorders) | 4 | 6
Pelvic hematoma (Blood and lymphatic system disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=60) | Treatment Arm (N=60)
Urinary tract infection (Infections and infestations) | 1 | 1
Acute urinary retention (Renal and urinary disorders) | 1 | 2
Small Bowel obstruction (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No